CLINICAL TRIAL: NCT02532504
Title: Change Your Life With Seven Sheets of Paper: A Pilot Randomized Controlled Trial for Postnatal Depression: A Pilot Randomized Controlled Trial for Postnatal Depression
Brief Title: Change Your Life With Seven Sheets of Paper
Acronym: CREATOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CREATOR001
Record Dates: First submitted 2015-08-15; First posted 2015-08-25 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2015-08

CONDITIONS: Postnatal Depression
Keywords: postnatal depression; Cognitive behaviour Therapy; Traditional Birth Attendants; low income country
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT seven sheets (Experimental): 8 sessions of CBT based intervention called "change your life with seven sheets of paper"
  Interventions: Other: CBT
- Treatment As Usual (No Intervention): Treatment As Usual

INTERVENTIONS:
Other: CBT — 8 sessions of CBT based intervention called "change your life with seven sheets of paper by Prof. Chris Williams. These sheets cover key skills of CBT that are;
  1. Five Areas vicious circle
  2. Bad thought spotter
  3. Amazing Bad thought Busting Programme (ABTPB)
  4. Easy 4 Step plan
  5. Things you do that mess you up/Confidence sheet
  6. Happy List/ Things you do that boost how you feel sheet
  7. Planner and Review sheets
  Arms: CBT seven sheets

SUMMARY:
The aim of this study is to deliver CBT based intervention called "Change your life with 7 Sheets of paper" to women with mild to moderate postnatal depression (PND) through trained traditional birth attendants (TBAs). Participants will be recruited from low income area in Karachi Pakistan. Edinburg Postnatal Depression scale (EPDS) will be used to screen mothers having children between birth till 12 months. Group intervention will be delivered through trained TBAs.

DETAILED DESCRIPTION:
The prevalence rate of PND in Pakistani women and its effect on the growth and development of young children and child mortality is very high. Despite availability of interventions to improve maternal health, the major issue in implementation of those interventions is because of limited availability of trained health professionals . Therefore the aim of this study is to train TBAs in delivering Cognitive Behaviour Therapy (CBT) based intervention called "Changing your life with seven sheets of paper". Participants will be recruited from low income area in Karachi. Total 36 participants will be recruited and randomized into 2 groups; intervention and Treatment As Usual (TAU) group. Total 8 sessions will be delivered by trained TBAs over the period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a child between 0-12 months
* Women who score 14 or above on Edinburgh Postnatal Depression scale (EPDS)
* Age range between 18 to 45 years
* Women able to provide written informed consent.

Exclusion Criteria:

* Severe depression or any other major psychiatric disorder
* Severe suicidal ideation
* Currently receiving any psychiatric or psychological treatment
* Intellectual disability in mother
* Chronic medical condition
* Having children with intellectual or physical disability

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Change in scores from baseline to 3rd month
  EPDS will be used to assess postnatal depression

SECONDARY OUTCOMES:
Patient health Questionnaire-9 | Change in scores from baseline to 3rd month
  PHQ-9 will be used to assess severity of depression
World Health Organization Quality of Life | Change in scoares from baseline to 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Batool Fatima, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Orangi Town, Karachi, Pakistan